CLINICAL TRIAL: NCT00551460
Title: S0535, A Phase II Study of ATRA, Arsenic Trioxide and Gemtuzumab Ozogamicin in Patients With Previously Untreated High-Risk Acute Promyelocytic Leukemia
Brief Title: S0535, Gemtuzumab and Combination Chemotherapy in Treating Patients With Previously Untreated Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0535; S0535 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Leukemia
Keywords: adult acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Gemtuzumab; Mercaptopurine; Methotrexate; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Induction:
  ATRA 45mg/m2 PO D1-CR Gemtuzumab Ozogamicin 9 mg/m2 IV D1 Arsenic Trioxide 0.15 mg/kg/d IV 5days/wk D10-CR
  Consolidation 1 and 2:
  Arsenic Trioxide 0.15 mg/kg/d IV 5days/wk x 5 weeks, repeat after 2 weeks rest
  Consolidation 2 and 3:
  ATRA 45 mg/m2 PO D1-7 Daunomycin 50 mg/m2/d IV D1-3
  Consolidation 5 and 6:
  GO 9mg/m2 IV D1
  Maintenance:
  ATRA 45 mg/m2/d PO D1-7 every 14 days 6-MP 60 mg/m2/d PO daily for 1 year Methotrexate 20 mg/m2 PO once/wk for 1 year
  Interventions: Drug: arsenic trioxide; Drug: gemtuzumab ozogamicin; Drug: mercaptopurine; Drug: methotrexate; Drug: tretinoin

INTERVENTIONS:
Drug: arsenic trioxide
Drug: gemtuzumab ozogamicin
Drug: mercaptopurine
Drug: methotrexate
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as gemtuzumab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Gemtuzumab may also stop the growth of promyelocytic leukemia by blocking blood flow to the cancer. Giving gemtuzumab together with combination chemotherapy may be more effective in treating promyelocytic leukemia.

PURPOSE: This phase II trial is studying how well giving gemtuzumab together with combination chemotherapy works in treating patients with previously untreated promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the event-free survival and death during the first six weeks in patients with previously untreated, high-risk acute promyelocytic leukemia treated with a combined regimen of tretinoin, arsenic trioxide, and gemtuzumab ozogamicin.
* To estimate the frequency and severity of toxicities of this regimen in this group of patients.
* To investigate the molecular response rate utilizing this regimen in high-risk patients.

OUTLINE:

* Induction chemotherapy: Patients receive oral tretinoin twice daily beginning on day 1 until CR (up to 90 days), gemtuzumab ozogamicin IV over 2 hours on day 1, and arsenic trioxide IV over 2 hours 5 days a week beginning on day 10 until CR (up to 60 days) in the absence of disease progression or unacceptable toxicity. Patients achieving A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status proceed to consolidation therapy after maintaining B1 peripheral blood status for ≥ 7 days.
* Consolidation therapy: Beginning between 2-8 weeks after documentation of complete response (CR), patients receive consolidation therapy.

  * Consolidation courses 1 and 2: Patients receive arsenic trioxide IV over 2 hours 5 days a week for 5 weeks. Treatment repeats every 7 weeks for up to 2 courses. Patients remaining in A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status continue with consolidation courses 3 and 4.
  * Consolidation courses 3 and 4: Within 4 weeks of completing consolidation course 2, patients receive oral tretinoin twice daily on days 1-7 and daunomycin IV bolus or over 1 hour on days 1-3. Within 2-8 weeks after recovery to B1 peripheral blood status, patients receive consolidation course 4 as in course 3. Patients who remain in B1 peripheral blood and C1 extramedullary disease status continue on consolidation courses 5 and 6.
  * Consolidation courses 5 and 6: Beginning between 2-8 weeks after recovery to B1 peripheral blood status, patients receive gemtuzumab IV over 2 hours on day 1. Between 2-8 weeks after recovery to B1 peripheral blood status, patients receive consolidation course 6 as in course 5. Patients who remain in A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status proceed to maintenance therapy.
* Maintenance therapy: Beginning 2-8 weeks after recovery of blood counts, patients receive oral tretinoin twice daily on days 1-7 every other week for 1 year, oral mercaptopurine once daily for 1 year, and oral methotrexate once weekly for 1 year.

Patients undergo bone marrow aspirates and biopsies periodically during study. Samples are analyzed for cytogenetics by fluorescence in situ hybridization (FISH) and for PML-RARα by polymerase chain reaction (PCR).

After completion of study treatment, patients are evaluated at 3, 6, 9, 12, 18, 24, and 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute promyelocytic leukemia (APL) based on bone marrow examination

  * APL-RARα-negative by RT-PCR are not eligible
* High-risk disease, defined as WBC > 100,000/mm^3
* Bone marrow specimens must be made available for cytogenetic studies

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prolonged QTc > 0.47 sec
* No other malignancy within the past 5 years, except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or stage II cancer from which the patients is currently in complete remission

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy for acute leukemia

  * At least 3 days since prior tretinoin (ATRA) allowed
* Prior hydroxyurea, corticosteroids, or leukapheresis to control high cell counts allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-11-15 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Lancet, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute; Rami Komrokji, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute; Cheryl L. Willman, MD, Study Chair — University of New Mexico Cancer Center; Marilyn L. Slovak, PhD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (192):
- United States (192):
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

REFERENCES:
- [Derived] Lancet JE, Moseley AB, Coutre SE, DeAngelo DJ, Othus M, Tallman MS, Litzow MR, Komrokji RS, Erba HP, Appelbaum FR. A phase 2 study of ATRA, arsenic trioxide, and gemtuzumab ozogamicin in patients with high-risk APL (SWOG 0535). Blood Adv. 2020 Apr 28;4(8):1683-1689. doi: 10.1182/bloodadvances.2019001278. PMID 32330241

RESULTS

PARTICIPANT FLOW:
Groups:
- ATRA + GO + Arsenic: Induction: ATRA 45mg/m2 PO D1-CR; Gemtuzumab Ozogamicin 9 mg/m2 IV D1; Arsenic Trioxide 0.15 mg/kg/d IV 5days/wk D10-CR
  Consolidation 1 and 2: Arsenic Trioxide 0.15 mg/kg/d IV 5days/wk x 5 weeks, repeat after 2 weeks rest
  Consolidation 2 and 3: ATRA 45 mg/m2 PO D1-7; Daunomycin 50 mg/m2/d IV D1-3
  Consolidation 5 and 6: GO 9mg/m2 IV D1
  Maintenance: ATRA 45 mg/m2/d PO D1-7 every 14 days; 6-MP 60 mg/m2/d PO daily for 1 year; Methotrexate 20 mg/m2 PO once/wk for 1 year
Period: Overall Study
Arm/Group | ATRA + GO + Arsenic
Started | 78
Completed | 60
Not Completed | 18
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Death | 7
Not completed — Ineligible | 4
Not completed — Not analyzable (did not start treatment) | 4

BASELINE CHARACTERISTICS:
Population: Baseline Participants includes eligible and analyzable patients. Ineligible patients and not analyzable patients from Participant Flow are excluded.
Arm/Group | ATRA + GO + Arsenic
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 46.5 [19.2 to 86.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 58
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Continuous Complete Remission at 3 Years
Description: Binary variable: yes if the patient achieves complete remission and remains in continuous complete remission until at least 3 years after entering the study; otherwise no.
Time Frame: 3 years
Population: The Analysis Population includes eligible and analyzable patients. Ineligible patients and not analyzable patients from Participant Flow are excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATRA + GO + Arsenic
Number analyzed (Participants) | 70
percentage of participants | 74 [62 to 84]

2. Primary Outcome: Mortality Rate at 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATRA + GO + Arsenic
Number analyzed (Participants) | 70
percentage of participants | 11 [5 to 21]

3. Secondary Outcome: Frequency of Toxicities
Description: Adverse events that were possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ATRA + GO + Arsenic
Number analyzed (Participants) | 70
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 37
  AST, SGOT | 46
  Acidosis (metabolic or respiratory) | 4
  Acute vascular leak syndrome | 1
  Adult respiratory distress syndrome (ARDS) | 3
  Albumin, serum-low (hypoalbuminemia) | 24
  Alkaline phosphatase | 23
  Alkalosis (metabolic or respiratory) | 4
  Allergic reaction/hypersensitivity | 8
  Allergic rhinitis | 6
  Allergy/Immunology-Other | 1
  Anorexia | 18
  Arthritis (non-septic) | 1
  Ascites (non-malignant) | 2
  Atelectasis | 2
  Atrioventricular block - 2nd degree Mobitz Type II | 1
  Atrioventricular block - first degree | 1
  Auditory/Ear-Other | 2
  Bicarbonate, serum-low | 7
  Bilirubin (hyperbilirubinemia) | 23
  Blood/Bone Marrow-Other | 4
  Bronchospasm, wheezing | 1
  Bruising (in absence of Gr 3-4 thrombocytopenia) | 8
  CNS cerebrovascular ischemia | 4
  Calcium, serum-high (hypercalcemia) | 1
  Calcium, serum-low (hypocalcemia) | 22
  Carbon monoxide diffusion capacity (DL(co)) | 1
  Cardiac Arrhythmia-Other | 1
  Cardiac General-Other | 2
  Cardiac troponin I (cTnI) | 1
  Cardiac troponin T (cTnT) | 1
  Cardiac-ischemia/infarction | 3
  Chelitis | 1
  Cholesterol, serum-high (hypercholesterolemia) | 4
  Confusion | 6
  Constipation | 26
  Cough | 17
  Creatinine | 5
  Cytokine release syndrome/acute infusion reaction | 1
  DIC (disseminated intravascular coagulation) | 19
  Dental: periodontal disease | 1
  Dermal change lymphedema, phlebolymphedema | 1
  Dermatology/Skin-Other | 3
  Diarrhea | 23
  Distention/bloating, abdominal | 10
  Dizziness | 4
  Dry mouth/salivary gland (xerostomia) | 1
  Dry skin | 11
  Dysphagia (difficulty swallowing) | 3
  Dyspnea (shortness of breath) | 27
  Edema, larynx | 1
  Edema: head and neck | 5
  Edema: limb | 33
  Edema: viscera | 2
  Encephalopathy | 1
  Esophagitis | 2
  Eyelid dysfunction | 1
  Fatigue (asthenia, lethargy, malaise) | 34
  Febrile neutropenia | 29
  Fever in absence of neutropenia, ANC lt1.0x10e9/L | 22
  Fibrinogen | 13
  Flatulence | 2
  Flushing | 2
  GGT (gamma-glutamyl transpeptidase) | 1
  Gastrointestinal-Other | 1
  Glomerular filtration rate | 2
  Glucose, serum-high (hyperglycemia) | 39
  Glucose, serum-low (hypoglycemia) | 1
  Hair loss/Alopecia (scalp or body) | 6
  Hearing: pts w/o audiogram not enroll monitor prgm | 1
  Heartburn/dyspepsia | 2
  Hematoma | 3
  Hemoglobin | 41
  Hemorrhage, Respiratory tract NOS | 3
  Hemorrhage, CNS | 8
  Hemorrhage, GI - Lower GI NOS | 2
  Hemorrhage, GI - Oral cavity | 4
  Hemorrhage, GI - Rectum | 1
  Hemorrhage, GI - Upper GI NOS | 2
  Hemorrhage, GU - Bladder | 1
  Hemorrhage, GU - Urinary NOS | 10
  Hemorrhage, GU - Vagina | 4
  Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS | 3
  Hemorrhage, pulmonary/upper respiratory - Lung | 1
  Hemorrhage, pulmonary/upper respiratory - Nose | 9
  Hemorrhage/Bleeding-Other | 8
  Hemorrhoids | 2
  Hepatobiliary/Pancreas-Other | 2
  Hiccoughs (hiccups, singultus) | 2
  Hot flashes/flushes | 1
  Hypertension | 25
  Hypotension | 4
  Hypoxia | 14
  INR (of prothrombin time) | 8
  Ileus, GI (functional obstruction of bowel) | 1
  Incontinence, anal | 1
  Induration/fibrosis (skin and subcutaneous tissue) | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Blood | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Colon | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Dental-tooth | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 4
  Inf (clin/microbio) w/Gr 3-4 neuts - Oral cav-gums | 3
  Inf (clin/microbio) w/Gr 3-4 neuts - Skin | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Stomach | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - Lung | 2
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 3
  Inf w/normal ANC or Gr 1-2 neutrophils - Up airway | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Vagina | 2
  Inf w/unknown ANC - Oral cavity-gums (gingivitis) | 1
  Infection (documented clinically or microbiologica | 1
  Infection with unknown ANC - Blood | 2
  Infection with unknown ANC - Lung (pneumonia) | 5
  Infection-Other | 1
  Injection site reaction/extravasation changes | 3
  Insomnia | 19
  Leak (including anastomotic), GU - Bladder | 1
  Left ventricular systolic dysfunction | 3
  Leukocytes (total WBC) | 26
  Liver dysfunction/failure (clinical) | 1
  Lymphopenia | 19
  Magnesium, serum-high (hypermagnesemia) | 16
  Magnesium, serum-low (hypomagnesemia) | 8
  Mental status | 1
  Metabolic/Laboratory-Other | 8
  Mood alteration - agitation | 3
  Mood alteration - anxiety | 14
  Mood alteration - depression | 10
  Mucositis/stomatitis (clinical exam) - Oral cavity | 2
  Mucositis/stomatitis (functional/symp) - Oral cav | 6
  Muscle weakness, not d/t neuropathy - Extrem-lower | 1
  Muscle weakness, not d/t neuropathy - body/general | 9
  Musculoskeletal/Soft Tissue-Other | 3
  Nasal cavity/paranasal sinus reactions | 3
  Nausea | 40
  Neurology-Other | 2
  Neuropathy: cranial - CN II Vision | 1
  Neuropathy: motor | 4
  Neuropathy: sensory | 3
  Neutrophils/granulocytes (ANC/AGC) | 38
  Obstruction, GU - Bladder | 1
  Ocular/Visual-Other | 5
  Optic disc edema | 2
  PTT (Partial thromboplastin time) | 13
  Pain - Abdomen NOS | 14
  Pain - Back | 8
  Pain - Bone | 2
  Pain - Buttock | 1
  Pain - Cardiac/heart | 1
  Pain - Chest/thorax NOS | 9
  Pain - Dental/teeth/peridontal | 1
  Pain - Esophagus | 2
  Pain - Extremity-limb | 5
  Pain - Eye | 2
  Pain - Face | 1
  Pain - Head/headache | 44
  Pain - Joint | 7
  Pain - Muscle | 7
  Pain - Neck | 3
  Pain - Oral cavity | 2
  Pain - Pleura | 1
  Pain - Sinus | 1
  Pain - Stomach | 1
  Pain - Throat/pharynx/larynx | 8
  Pain - Urethra | 2
  Pain-Other | 6
  Petechiae/purpura (hemorrhage into skin or mucosa) | 15
  Phosphate, serum-low (hypophosphatemia) | 7
  Platelets | 40
  Pleural effusion (non-malignant) | 9
  Pneumonitis/pulmonary infiltrates | 3
  Potassium, serum-high (hyperkalemia) | 9
  Potassium, serum-low (hypokalemia) | 28
  Prolonged QTc interval | 21
  Proteinuria | 6
  Pruritus/itching | 12
  Psychosis (hallucinations/delusions) | 1
  Pulmonary/Upper Respiratory-Other | 5
  Rash/desquamation | 26
  Renal failure | 4
  Renal/Genitourinary-Other | 2
  Retinoic acid syndrome | 6
  Rigors/chills | 7
  SVT and nodal arrhythmia - Atrial fibrillation | 1
  SVT and nodal arrhythmia - SVT arrhythmia NOS | 1
  SVT and nodal arrhythmia - Sinus arrhythmia | 3
  SVT and nodal arrhythmia - Sinus bradycardia | 5
  SVT and nodal arrhythmia - Sinus tachycardia | 20
  Seizure | 1
  Sodium, serum-high (hypernatremia) | 5
  Sodium, serum-low (hyponatremia) | 19
  Soft tissue necrosis - Extremity-lower | 1
  Somnolence/depressed level of consciousness | 6
  Speech impairment (e.g., dysphasia or aphasia) | 1
  Stricture/stenosis (incl anastomotic) GI - Pharynx | 1
  Sweating (diaphoresis) | 9
  Syncope (fainting) | 2
  Syndromes-Other | 4
  Taste alteration (dysgeusia) | 2
  Thrombosis/embolism (vascular access-related) | 1
  Thrombosis/thrombus/embolism | 2
  Thyroid function, low (hypothyroidism) | 1
  Triglyceride, serum-high (hypertriglyceridemia) | 11
  Ulceration | 2
  Uric acid, serum-high (hyperuricemia) | 2
  Urinary frequency/urgency | 1
  Urinary retention (including neurogenic bladder) | 4
  Urine color change | 1
  Vaginal discharge (non-infectious) | 1
  Ventricular arrhythmia - PVCs | 1
  Ventricular arrhythmia - Ventricular tachycardia | 1
  Vision-blurred vision | 7
  Vision-flashing lights/floaters | 2
  Vision-photophobia | 4
  Vitreous hemorrhage | 3
  Voice changes/dysarthria | 1
  Vomiting | 33
  Watery eye (epiphora, tearing) | 2
  Weight gain | 3
  Weight loss | 9

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Only adverse events and serious adverse events that are possibly, probably or definitely related to study drug are reported.
Groups:
- ATRA + GO + Arsenic: Induction: ATRA 45mg/m2 PO D1-CR; Gemtuzumab Ozogamicin 9 mg/m2 IV D1; Arsenic Trioxide 0.15 mg/kg/d IV 5days/wk D10-CR
Arm/Group | ATRA + GO + Arsenic
All-Cause Mortality (participants affected / at risk) | 10/70
Serious Adverse Events (participants affected / at risk) | 11/70
Other Adverse Events (participants affected / at risk) | 68/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATRA + GO + Arsenic (N=70)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac General-Other (Cardiac disorders) | 1
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1
Infection with unknown ANC - Blood (Infections and infestations) | 2
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT (Investigations) | 2
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1
Leukocytes (total WBC) (Investigations) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Platelets (Investigations) | 3
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 1
Renal/Genitourinary-Other (Renal and urinary disorders) | 2
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmo/upper resp- Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 1
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATRA + GO + Arsenic (N=70)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 4
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 29
Hemoglobin (Blood and lymphatic system disorders) | 40
SVT and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 5
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 19
Ocular/Visual-Other (Eye disorders) | 5
Vision-blurred vision (Eye disorders) | 7
Vision-photophobia (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 26
Diarrhea (Gastrointestinal disorders) | 23
Distention/bloating, abdominal (Gastrointestinal disorders) | 10
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 40
Pain - Abdomen NOS (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 33
Edema: head and neck (General disorders) | 5
Edema: limb (General disorders) | 33
Fatigue (asthenia, lethargy, malaise) (General disorders) | 34
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 22
Pain - Chest/thorax NOS (General disorders) | 9
Pain-Other (General disorders) | 6
Rigors/chills (General disorders) | 7
Syndromes-Other (General disorders) | 4
Allergic reaction/hypersensitivity (Immune system disorders) | 8
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 4
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 8
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 36
AST, SGOT (Investigations) | 44
Alkaline phosphatase (Investigations) | 23
Bilirubin (hyperbilirubinemia) (Investigations) | 22
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 4
Creatinine (Investigations) | 5
Fibrinogen (Investigations) | 13
INR (of prothrombin time) (Investigations) | 8
Leukocytes (total WBC) (Investigations) | 25
Lymphopenia (Investigations) | 19
Metabolic/Laboratory-Other (Investigations) | 8
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 37
PTT (Partial thromboplastin time) (Investigations) | 13
Platelets (Investigations) | 37
Prolonged QTc interval (Investigations) | 21
Weight loss (Investigations) | 9
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 24
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 18
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 7
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 22
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 39
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 16
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 9
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 28
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 5
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 19
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 11
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 9
Pain - Back (Musculoskeletal and connective tissue disorders) | 8
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain - Joint (Musculoskeletal and connective tissue disorders) | 7
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 4
Hemorrhage, CNS (Nervous system disorders) | 7
Neuropathy: motor (Nervous system disorders) | 4
Ocular/Visual-Other (Nervous system disorders) | 5
Pain - Head/headache (Nervous system disorders) | 44
Somnolence/depressed level of consciousness (Nervous system disorders) | 5
Confusion (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 19
Mood alteration - anxiety (Psychiatric disorders) | 14
Mood alteration - depression (Psychiatric disorders) | 10
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 10
Proteinuria (Renal and urinary disorders) | 6
Renal failure (Renal and urinary disorders) | 4
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 4
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 26
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 5
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 11
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 6
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 15
Pruritus/itching (Skin and subcutaneous tissue disorders) | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 26
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 9
Hemorrhage/Bleeding-Other (Vascular disorders) | 8
Hypertension (Vascular disorders) | 24
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT00551460/Prot_SAP_ICF_000.pdf